CLINICAL TRIAL: NCT02756117
Title: The Effect of Acute Lysine Administration on α-aminoadipic Acid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Jane Ferguson, Principal Investigator, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 160520
Record Dates: First submitted 2016-04-25; First posted 2016-04-29 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Healthy; Pre-diabetic
MeSH Terms: conditions — Glucose Intolerance | interventions — Lysine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy (Experimental): 10 Healthy subjects will be enrolled and each will undergo study procedures at one study visit. After screening and consent have been conducted over the phone, subjects will participate in the study procedures. Subjects will arrive in a fasting state (no eat or drink for 8 hours, excluding water). Following collection of blood pressure, height, weight, and a urine and blood sample, subjects will be given an oral bolus of L-lysine (10 g) in 100 ml water. This amount of lysine is equivalent to that which is found in a 10oz. serving of beef. Subjects will provide additional urine and blood samples serially post-ingestion. Because blood draws will be collected through an IV, Normal (0.9%) Saline (NS) will be infused at a rate of 10 ml/hr to flush the canula prior to each blood draw.
  All subjects will undergo the same procedures and interventions.
  Interventions: Drug: L-Lysine; Drug: Normal (0.9%) Saline

INTERVENTIONS:
Drug: L-Lysine
Drug: Normal (0.9%) Saline
  Other Names: NS

SUMMARY:
This study aims to assess the effect and breakdown of lysine administration, specifically examining whether it leads to increased plasma 2-AAA in healthy humans.

DETAILED DESCRIPTION:
The significance of diabetes and related co-morbidities as considerable health concerns in the US and worldwide is clearly supported by the high incidence (estimated 9.3% of the US population), mortality burden (7th leading cause of death in the US), and rising costs ($245 billion/year). Strategies to identify individuals at high diabetic risk, and to modulate disease processes in these individuals before the onset of overt disease, would have a significant impact in reducing mortality, morbidity and healthcare costs. For this approach to be successful, early markers of disease that predict at-risk individuals before onset of dysregulated glycemic control are required, as well as discovering novel pathways for therapeutic targeting.

The purpose of this study is to investigate a novel biomarker, α-aminoadipic acid (2-AAA), which may influence the risk of diabetes. 2-AAA has been identified as a novel predictor of diabetes development in humans, identifying at-risk individuals before any detectable glucose abnormalities. 2-AAA is a naturally occurring metabolite in the body, and it has no known adverse effects at normal physiological levels. 2-AAA is generated in the body from the breakdown of lysine. Lysine is one of the twenty essential amino acids, meaning that it is essential for human function, but that our body cannot manufacture it. Thus, it is acquired from dietary sources (such as meat, eggs, soybeans and legumes), with a recommended daily intake of 30 mg/kg/day. Amino acids are the building blocks of proteins, which are what allow our cells, organs and body to maintain structure and function. The investigators are interested in whether 2-AAA is increased in the body after consumption of lysine.

The investigators specific aim is to determine whether acute lysine administration leads to increased plasma 2-AAA in humans. Catabolism of lysine leads to generation of 2-AAA. In this study, the investigators will determine whether a single dose of lysine leads to increased plasma 2-AAA present in the blood and urine of humans. The investigators will ask 10 lean, healthy subjects to drink a beverage containing lysine and the investigators will measure the level of 2-AAA in their blood plasma and urine at baseline (before ingestion) and serially post-ingestion. The amount of lysine subjects will be given is equivalent to that which is found in a 10 oz. serving of beef. This pilot study will allow us to establish the relationship between lysine and 2-AAA in healthy subjects, and inform future studies on how to study the effects of 2-AAA on diabetes risk.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18 to <25 kg/m2
* Men and women ages 18-45 years

Exclusion Criteria:

* Current use of prescription medications (apart from hormonal birth control)
* Current use of amino acid supplements (including branched-chain amino acids) or supplemental protein (habitual consumption of protein powder, bars, shakes), and unwilling to temporarily discontinue use (1 week prior to study visit)
* Individuals who currently use tobacco products or have done so in the previous 30 days
* Prior or current cardiovascular disease, renal disease, or liver disease
* Diabetes mellitus (taking insulin, other anti-diabetic agents, or diet-controlled)
* Atrial fibrillation
* Bleeding disorder or anemia
* Positive pregnancy test
* Women who are breastfeeding
* Participation in another clinical trial within the previous 6 weeks prior to the study visit
* Inability to provide written informed consent
* Inability to fast for 8 hours

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Change in plasma 2-AAA from baseline to peak post-lysine ingestion (anticipated 2-4 hours post-ingestion) | Baseline and 2-4 hours
  The primary goal is to detect whether there is a measurable increase in 2-AAA in plasma following lysine administration. Samples will be measured at baseline (pre-ingestion) and serially post-ingestion. Relative concentrations are determined through mass spectrometry, and expressed in arbitrary units.

SECONDARY OUTCOMES:
Change in urinary 2-AAA from baseline to peak post-lysine ingestion (anticipated 2-4 hours post-ingestion) | Baseline and 2-4 hours
  A secondary goal is to detect whether there is a measurable increase in 2-AAA in urine following lysine ingestion. Relative concentrations are determined through mass spectrometry, and expressed in arbitrary units.

CONTACTS AND LOCATIONS:
Overall Officials: Jane F Ferguson, PhD, Principal Investigator — Vanderbilt Cardiovascular Medicine

IPD SHARING:
Plan to Share IPD: Yes